CLINICAL TRIAL: NCT06037577
Title: A Double-Blind, Randomized, Placebo-Controlled, Phase I Study To Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Escalating Subcutaneous Doses of CM-101 in Healthy Male Subjects
Brief Title: Subcutaneous Doses of CM-101 as a Treatment for Medical Conditions Involving Inflammatory and Fibrotic Mechanisms in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ChemomAb Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CM-101-SC-001
Record Dates: First submitted 2023-08-30; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Nonalcoholic Steatohepatitis (NASH); Primary Sclerosing Cholangitis (PSC); Systemic Sclerosis (SSc)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Cholangitis, Sclerosing; Scleroderma, Systemic | interventions — streptococcal polysaccharide type III group B

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti-human CCL24 monoclonal antibody (CM-101) (Experimental): Single 5 mg/kg of CM-101, Subcutaneous administration
  Interventions: Drug: CM-101
- Placebo (Placebo Comparator): Placebo : Subcutaneous administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CM-101 — Anti-human CCL24 monoclonal antibody (CM-101)
  Arms: Anti-human CCL24 monoclonal antibody (CM-101)
Drug: Placebo — Placebo Comparator
  Arms: Placebo

SUMMARY:
CM-101 is developed as treatment for medical conditions involving inflammatory and fibrotic mechanisms such as non-alcoholic steatohepatitis (NASH) and primary sclerosing cholangitis (PSC) and systemic sclerosis (SSc). In this current study, the IP is tested in healthy male volunteers.

DETAILED DESCRIPTION:
A single-center, randomized double-blind, placebo-controlled, single-dose study Healthy volunteers were screened for up to 28 days prior to drug administration. The study included one dose group of 8 subjects. A single 5 mg/kg CM-101 dose was subcutaneously administered. The study was comprised of a screening period, a treatment day, a follow-up (FU) period of 42 days and an end of study (EOS) FU visit.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must provide written informed consent prior to participating in the study.
2. Considered healthy by the Investigator as defined by no clinically relevant abnormalities identified by a detailed medical history, full physical examination, 12-lead ECG, and clinical laboratory tests.
3. Body Mass Index (BMI) 19.0-29.0 kg/m2 and total body weight within 55-95 Kg.
4. Fertile men must agree to use a barrier contraceptive (condom) for 90 days post-dosing and are restricted from donating sperm for 90 days after dosing. Subjects with a vasectomy performed more than 6 months prior to treatment are also acceptable.
5. Non-smoking and no use of any tobacco or nicotine product by declaration for a period of at least 3 months prior to screening.
6. Supine blood pressure and heart rate within normal limits (systolic 90-140 mmHg; diastolic 50-90 mmHg, heart rate 45-100 beats per minute). No evidence of orthostatic hypotension.
7. ECG with no clinically significant abnormalities recorded at Screening visit and on dosing day (before drug administration): PR interval within 120 and 210 ms, QRS interval< 120 ms, and QTc interval <450 ms.
8. Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Evidence or history of clinically relevant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies,). This includes any acute or chronic medical or psychiatric condition or laboratory abnormality.
2. History or current drug/alcohol abuse. History of regular alcohol consumption exceeding - 14 drinks/week for men (1 drink = 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within 6 months of screening.
3. Hypereosinophilia defined as peripheral blood Eosinophils > 4.5×108/L (450/μl) or exceeding 7% of the circulating leukocytes.
4. Positive urine drugs of abuse (DoA) test during screening and on admission.
5. Positive breath alcohol test on admission.
6. Known acute or chronic allergy to any drug or hypersensitivity to any of the test formulation compounds or contraindication to the test product.
7. Use of any prescription or over-the-counter (OTC) medications, including vitamins and herbal or dietary supplements within 14 days prior to dosing. Paracetamol for symptomatic relief of pain is allowed up to 24 hours prior to study drug administration.
8. Having received any biological treatment with recombinant antibodies, immunological therapy, or anticancer treatment. Previous standard vaccination treatment is allowed.
9. Positive HIV, hepatitis HBsAg or hepatitis HCV Ab serology tests at Screening.
10. Subjects who donated blood in the 3 months or received blood or plasma derivatives in the 6 months preceding study drug administration.
11. Participation in another clinical trial within 3 months prior to dosing (calculated from the previous study's last dosing day).
12. Subjects with any acute medical situation (e.g. acute infection) within 48 hours of dosing.
13. Subjects with an inability to communicate well with the investigators and CRC staff (e.g., language problem, poor mental development).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy Male Subjects
Enrollment: 8 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2019-05-05 (Actual); Study Completion 2019-05-05 (Actual)

PRIMARY OUTCOMES:
Incidence and characteristics of adverse events (AEs) | 10 weeks
  Incidence and characteristics of adverse events (AEs) occurring following single subcutaneous doses of CM-101
Plasma pharmacokinetic (PK) of CM-101 - Maximum CM-101 plasma concentration (Cmax) | 10 weeks
  Maximum CM-101 plasma concentration (Cmax)
Plasma pharmacokinetic (PK) of CM-101 - Time to Cmax (tmax) | 10 weeks
  Time to Cmax (tmax)
Plasma pharmacokinetic (PK) of CM-101 - Area under the curve (AUC) to the final concentration ≥ limit of quantitation (LOQ), AUC(0-t) and to infinity AUCinf | 10 weeks
  Area under the curve (AUC) to the final concentration ≥ limit of quantitation (LOQ), AUC(0-t) and to infinity AUCinf
Plasma pharmacokinetic (PK) of CM-101 - Terminal elimination rate constant (λz) | 10 weeks
  Terminal elimination rate constant (λz)
Plasma pharmacokinetic (PK) of CM-101 - Terminal elimination half-life (T½) | 10 weeks
  Terminal elimination half-life (T½)

SECONDARY OUTCOMES:
Assessment, based on the safety profile within the tested doses range of CM-101 - dose-limiting toxicity (DLT) | 10 weeks
  Assessment, based on the safety profile, whether dose-limiting toxicity (DLT) is attained within the tested doses range of CM-101
Assessment, based on the safety profile within the tested doses range of CM-101 - maximum tolerated dose (MTD) | 10 weeks
  Assessment, based on the safety profile, whether maximum tolerated dose (MTD) is attained within the tested doses range of CM-101
Level of antibodies | 10 weeks
  Level of antibodies against CM-101

CONTACTS AND LOCATIONS:
Overall Officials: Arnon Aharon, MD, Study Director — ChemomAb Ltd.
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel